CLINICAL TRIAL: NCT02344550
Title: Ovarian Suppression Plus Letrozole Plus Everolimus for Hormone Receptor-Positive, Tamoxifen and Ovarian Suppression Pretreated, Premenopausal Women With Recurrent or Metastatic Breast Cancer[LEO]
Brief Title: Study of GnRH-A [Leuprorelin(Lorelin Depot] Plus Leterozole +/- Everolimus for Premenopausal Women With Metastatic Breast Cancer
Acronym: LEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Bae Kim, M.D., Ph D., Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2013-0720; AMC (Other: Asan Medical Center)
Record Dates: First submitted 2014-05-07; First posted 2015-01-26 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; HER2 negative; hormone-receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Letrozole; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus arm (Experimental): Everolimus 10mg p.o. daily Letrozole 2.5 mg p.o. daily Leuprorelin (Leuprolide) 3.75mg SC every 4 weeks
  Interventions: Drug: Everolimus(afinitor); Drug: Letrozole; Drug: Leuprolide(Lorelin Depot)
- Control arm (Active Comparator): Letrozole 2.5 mg p.o. daily Leuprorelin (Leuprolide) 3.75mg SC every 4 weeks
  Interventions: Drug: Letrozole; Drug: Leuprolide(Lorelin Depot)

INTERVENTIONS:
Drug: Everolimus(afinitor) — Everolimus 10mg p.o. daily
  Other Names: Afinitor
  Arms: Everolimus arm
Drug: Letrozole — Letrozole 2.5 mg p.o. daily
  Other Names: Femara
Drug: Leuprolide(Lorelin Depot) — Leuprorelin (Lorelin Depot)3.75 mg SC in every 4 weeks
  Other Names: Leuprorelin (Dongkook Pharm Co Ltd)

SUMMARY:
The purpose of this study is to evaluate the efficacy of addition of everolimus to letrozole with LHRH agonist in premenopausal metastatic breast cancer patients who failed to tamoxifen treatment.

DETAILED DESCRIPTION:
Endocrine therapy is the cornerstone of treatment for patients with hormone receptor (HR)-positive advanced breast cancer. The selection of endocrine agents takes account of the menopausal status, the type of previous adjuvant endocrine treatment, the disease free interval and past medical history1.

The goal of endocrine treatment is to block or interfere with the function of estrogen or progesterone. The major source of estrogen in premenopausal women is the ovaries. In premenopausal women with HR-positive advanced breast cancer, tamoxifen, ovarian function suppression or a combination of those have been used. Unfortunately, not all patients have a response to first-line endocrine therapy, and even patients who have a response will eventually become resistant. Patients experiencing disease progression with a first-line endocrine therapy may benefit from other endocrine agents, such as aromatase inhibitors (steroidal or nonsteroidal) and the estrogen receptor (ER) antagonist2-5. Aromatase inhibitors combined with luteinizing hormone-releasing hormone (LHRH) analogs or ovarian ablation are also a feasible treatment modality for premenopausal patients with HR-positive advanced breast cancer6.

An emerging mechanism of endocrine resistance in aberrant signaling through the phosphatidylinositol 3-kinase (PI3K)-Akt-mammalian target of rapamycin (mTOR) signaling pathway7-9. Growing evidence supports a close interaction between the mTOR pathway and ER signaling. A substrate of mTOR complex 1 (mTORC1), called S6 kinase 1, phosphorylates the activation function domain 1 of ER, which is responsible for ligand-independent receptor activation10. Everolimus is a sirolimus derivative that inhibits mTOR through allosteric binding to mTORC111. In preclinical models, the use of everolimus in combination with aromatase inhibitors results in synergistic inhibition of the proliferation and induction of apoptosis12. In a randomized, phase 2 study comparing neoadjuvant everolimus plus letrozole with letrozole alone in patients with newly diagnosed ER-positive breast cancer, the response rate for the combination was higher than that for letrozole alone13. Recently, the Breast Cancer Trials of Oral Everolimus-2 (BOLERO-2) study showed that the addition of everolimus to exemestane significantly improved progression-free survival, with observed medians of 6.9 and 2.8 months, corresponding to a 57% reduction in the hazard ratio14.

Based on this rationale, the investigators introduced randomized trial to evaluate the efficacy of addition of everolimus to letrozole with LHRH agonist in premenopausal metastatic breast cancer patients who failed to tamoxifen treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Histologically or cytologically confirmed, HER-2 negative breast cancer with recurrent or metastatic disease
* No HER2 overexpressing breast cancer
* Premenopausal status, defined as either
* ER and/or PR positive
* Progressive disease on tamoxifen treatment or sequential or combined treatment of tamoxifen and GnRH agonist as a palliative or an adjuvant endocrine treatment
* Duration of tamoxifen treatment should be at least 3 months or more
* No prior treatment with an aromatase inhibitor or inactivator or fulvestrant, or mTOR inhibitors
* One line of chemotherapy in metastatic setting is permitted
* ECOG performance status 0,1 or 2
* At least one measurable lesion or mainly lytic bone lesions in the absence of measurable disease
* Adequate hematologic, liver and kidney function

Exclusion Criteria:

* Pregnant women or patients in lactation
* More than one line of prior chemotherapy for metastatic breast cancer
* GnRH agonist with tamoxifen treatment within 2 weeks.
* Active malignancy other than breast cancer, in situ carcinoma of the cervix, controlled resected thyroid well differentiated carcinoma or non-melanomatous skin cancer in the past 5 years
* Active cardiovascular disease such as angina, ventricular tachycardia, uncontrolled hypertension
* Active uncontrolled infection
* Symptomatic brain metastases
* Lymphangitic carcinomatosis involving >50% of the lungs
* Evidence of metastases involving more than one third of the liver on sonogram or CT
* Patients not able or unwilling to give informed consent

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Participants will be followed every 8 weeks , up to 12 Months
  At time disease progression

SECONDARY OUTCOMES:
Overall Response rate | Participants will be followed every 8 weeks, up to 12 Months
  At time disease evaluation

OTHER OUTCOMES:
Clinical benefit rate (CBR) | Participants will be followed every 8 weeks, up to 12 Months
  At time disease progression
Overall survival | Participants will be followed every 8 weeks, up to 12 Months
  At time of death occur or follow-up loss
Number of patients with adverse events | Participants will be followed every 8 weeks, up to 12 Months
  During treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bae Kim, M.D., Ph D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea